CLINICAL TRIAL: NCT04322461
Title: Effect of Exercise, Endocannabinoids and Ketones on Cerebral Metabolism in a Cognitive Disorders Population : Pilot Project PARKA
Brief Title: Effect of Exercise, Endocannabinoids and Ketones on Cerebral Metabolism in a Cognitive Disorders Population
Acronym: PARKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-3436
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Parkinson Disease; Alzheimer Disease
Keywords: Alzheimer; Parkinson; Ketones; medium chain triglycerides; cognition; brain
MeSH Terms: conditions — Parkinson Disease; Alzheimer Disease; Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson disease (Experimental): 2 months intervention with 50g/day of a commercial MCT supplement combine with supervised aerobic exercise 3x/week.
  Interventions: Dietary Supplement: Betaquik MCT supplement
- Alzheimer's disease (Experimental): 2 months intervention with 50g/day of a commercial MCT supplement combine with supervised aerobic exercise 3x/week.
  Interventions: Dietary Supplement: Betaquik MCT supplement

INTERVENTIONS:
Dietary Supplement: Betaquik MCT supplement — 50g/day divided in 3. Breakfast, lunch and dinner

SUMMARY:
A two months intervention in which two groups of cognitive disorders, Parkinson and Alzheimer's disease, will receive 50g/day of a commercial MCT supplement combined with supervised aerobic exercise 3 times/week. Cognition and ketones will be assess before and after the intervention, along with endocannabinoids plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's or parkinson disease diagnostic
* Stable medication associated with the disease
* Able to consent
* Presence of an accompanying person for the first and last visit.
* Ability to read and talk in French

Exclusion Criteria:

* MMSE < 20
* MCT or coconut oil supplementation
* Coconut allergy
* Cannabis, THC or CBD consumption
* Excessive alcohol consumption
* Physical activity 3x/week
* Presence of an metallic object in the body
* Impossibility to lay in dorsal decubitus for 40 minutes
* Cardiac disease
* Any uncontrolled disease that could interfer with the project.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Cognition | 2 months, evaluation before and after intervention
  Measure of cognition with CANTAB
Ketones | 2 months, evaluation before and after intervention
  Measurement of ketones concentrations

SECONDARY OUTCOMES:
Endocannabinoids | 2 months, evaluation before and after intervention
  Endocannabinoids plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No